CLINICAL TRIAL: NCT01574599
Title: A Randomized Controlled Evaluation of a Repetitive Facilitative Exercise Program for Adults With an Established Stroke and Upper Extremity Impairment
Brief Title: Use of Repetitive Facilitative Exercise Program in Established Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor subject recruitment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Billie A. Schultz, MD; Consultant in Department of Physical Medicine and Rehabilitation, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 11-005596
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Stroke
Keywords: Stroke; weakness; rehabilitation; chronic stroke
MeSH Terms: conditions — Stroke; Asthenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Repetitive Facilitative Exercise (Experimental): Occupational therapy program - Repetitive facilitative exercise therapy protocol including 40 min of RFE and 20 minutes of task-specific activity. 3 treatment sessions weekly for a total of 4 weeks.
  Interventions: Other: Occupational therapy- Repetitive Facilitative Exercise
- Conventional Therapy Program (No Intervention): Typical therapy excluding robotics, RFE

INTERVENTIONS:
Other: Occupational therapy- Repetitive Facilitative Exercise — Occupational therapy program - Repetitive facilitative exercise therapy protocol including 40 min of RFE and 20 minutes of task-specific activity. 3 treatment sessions weekly for a total of 4 weeks.
  Arms: Repetitive Facilitative Exercise

SUMMARY:
The purpose of this study is to assess whether a novel therapy approach (repetitive facilitative exercise (RFE)) is more effective than conventional rehabilitation in facilitating the recovery of upper extremity function following stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Having a single ischemic or hemorrhagic hemispheric stroke of more than 6 months duration
* The ability to selectively demonstrate active extension of at least 10 degrees at the metacarpo-phalangeal joint and the interphalangeal joints and 20 degrees at the wrist
* Capable of effectively participating in the study

Exclusion Criteria:

* Upper extremity contracture/pain that interfere with study technique
* Pre-existing upper extremity neurologic or orthopedic disorders
* Unstable medical condition
* BMI > 35
* Active treatment of condition during 3 months prior to enrollment in study (botulinum toxin, therapy, tendon release, etc.)
* Language or cognitive/perceptual deficits or scheduling problems that would limit participation
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Arm score | baseline, immediate post-intervention and 3 month post-intervention

SECONDARY OUTCOMES:
Motor Activity Log | baseline, immediate post-intervention and 3 month post-intervention
9-Hole Peg Test | baseline, immediate post-intervention and 3 month post-intervention
Box and Block test | baseline, immediate post-intervention and 3 month post-intervention
Grasp strength | baseline, immediate post-intervention and 3 month post-intervention
Active Range of motion of shoulder flexion, wrist extension, and index finger extension | baseline, immediate post-intervention and 3 month post-intervention
Overall patient satisfaction | baseline, immediate post-intervention and 3 month post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Billie Schultz, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States